CLINICAL TRIAL: NCT05437068
Title: Effects of Oral Nutritional Supplementation in 12-71 Months Old Children at Risk of Undernutrition
Brief Title: Nutritional Supplementation in Children at Risk of Undernutrition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research focus
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL55
Record Dates: First submitted 2022-06-15; First posted 2022-06-29 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Nutritional Supplement (ONS) Group (Experimental): Two servings per day in addition to dietary counseling
  Interventions: Other: Oral Nutritional Supplement (ONS)

INTERVENTIONS:
Other: Oral Nutritional Supplement (ONS) — ONS plus dietary counseling

SUMMARY:
This is a prospective, multicenter, single-arm intervention study. The expected duration of study participation for each participant is approximately 120 days. The current study aims to investigate the effectiveness of an ONS formula in children at risk or with undernutrition in Thailand.

ELIGIBILITY:
Inclusion Criteria:

Child is between 1 year 0 days to 5 years 364 days old at enrolment

Undernourished or at risk of undernutrition, defined as:

* WHZ <- 1 and HAZ <-1 for children up to 4 years 364 days, according to the WHO Growth Standards; or
* BMIAZ <-1 and HAZ <-1 for children 5 years 0 days and older, according to the WHO Growth Reference Standards

Child is not currently breastfed

Child's parent(s)/LG is willing to abstain from giving additional non-study Oral Nutritional Supplement (ONS) other than the study product during the study intervention period

Child is a singleton

Child's parent(s)/LG is able and willing to follow study procedures and record data in parent diary and complete any forms or assessments needed throughout the study

Child's parent(s)/LG is not planning to relocate during the study period

Child's parent(s)/LG has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) or other applicable privacy regulation authorization prior to any participation in the study

Exclusion Criteria:

Child participates in another study that has not been approved as a concomitant study

Child is known to have galactosemia, be allergic or intolerant to any ingredient found in the study product

Child had a history of preterm delivery, defined as a birth before 37 completed weeks of gestation as reported by parent(s)/LG

Child had birth weight < 2500 g or > 4000 g

Child whose either parent has BMI ≥ 27.5 kg/m2

Child has current acute or chronic infections including but not restricted to respiratory infections, diarrhea, acute and chronic Hepatitis B or C, HIV infection or tuberculosis

Child has been diagnosed with the following:

* Severe gastrointestinal disorders such as celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic fibrosis
* Neoplastic, renal, hepatic or cardiovascular, hormonal or metabolic disorders, congenital disease or genetic disorders such as atrial or ventricular wall defects, Down's syndrome, or thalassemia
* Infantile anorexia nervosa, developmental disability, including physical disorders such as cerebral palsy, or developmental delay
* Disorders of hemoglobin structure, function or synthesis

Clinically significant nutritional deficiency requiring specific treatment with another nutritional supplement (other than the study product)

Any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Height-for-age-Z-score | Baseline to 120 days
  Change in Height-for-age-Z-score

SECONDARY OUTCOMES:
Weight | Baseline to 30 days and 120 days
  Measured in Kg
Height | Baseline to 30 days and 120 days
  Measured in cm
Mid-Upper-Arm Circumference (MUAC) | Baseline to 30 days and 120 days
  Measured in cm
Weight-for-Height Measurement Calculations | Baseline to 30 days and 120 days
  Weight-for-height standard z scores and percentiles
Weight-for-Age Measurement Calculations | Baseline to 30 days and 120 days
  Weight-for-age standard z scores and percentiles
BMI-for-Age Measurement Calculations | Baseline to 30 days and 120 days
  BMI-for-age standard z scores and percentiles
Height-for-Age Measurement Calculations | Baseline to 30 days and 120 days
  Height-for-age standard z scores and percentiles
MUAC-for-Age Measurement Calculations | Baseline to 30 days and 120 days
  MUAC-for-age standard z scores and percentiles
Dietary Intake | Baseline to 30 days and 120 days
  Measured by 24-hour dietary recall
Appetite | Baseline to 30 days and 120 days
  Visual analog scale from 0 (Ate Very Little) to 10 (Ate Very Much) with high scores being favorable
Physical Activity | Baseline to 30 days and120 days
  Visual analog scale from 0 (Not Active) to 10 (Very Active) with high scores being favorable

OTHER OUTCOMES:
Parental Evaluation of Child's Healthy Growth | Baseline to 30 days and 120 days
  Parent-reported satisfaction and assessment of child's healthy growth on 10-point visual analog scale, scored from 0 Very dissatisfied/Strongly disagree to 10 Very satisfied/Strongly agree, with higher scores being favorable
Parental Assessment of Child's Sleep | Baseline to 30 days and 120 days
  Parent-reported questionnaire of child's usual amount of sleep (hours and minutes), and number (number of times) and length (minutes) of awakenings per night
Adverse Event | Baseline to 120 days
  Number of participants with reported adverse events
Illness Questionnaire | Baseline to 120 days
  Parent reported number of sick episodes, sick days, healthcare visits and symptoms, with higher number reported being less favorable
Mid Upper Arm Muscle Circumference (MUAMC) Calculation | Baseline to 30 days and 120 days
  Changes in MUAMC calculations
Arm Muscle Area (AMA) Calculation | Baseline to 30 days and 120 days
  Changes in AMA calculations
Arm Fat Area (AFA) Calculation | Baseline to 30 days and 120 days
  Changes in AFA calculations
Arm Fat Index (AFI) Calculation | Baseline to 30 days and 120 days
  Changes in AFI calculations

CONTACTS AND LOCATIONS:
Overall Officials: Yen Ling Mandy Ow, PhD, Study Chair — Abbott Nutrition

IPD SHARING:
Plan to Share IPD: No